CLINICAL TRIAL: NCT02116283
Title: Mobile Sensing of Smoking Behavior
Acronym: Mobi-Smoke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00044941
Record Dates: First submitted 2014-01-16; First posted 2014-04-16 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-11

CONDITIONS: Smoking; Health
Keywords: smoking; healthy; smartphone
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: 48 hour smoking abstinence — Participants will maintain smoking abstinence for 48 hours
Other: Smartphone — Participants will use an Android-based smartphone as their own for one month

SUMMARY:
Smokers will use a smartphone app on a smartphone provided for the study that will passively sense and record information about their activities. Information collected from the smartphone app will be used to develop future smartphone apps that will predict when an individual is at risk of smoking.

DETAILED DESCRIPTION:
Smokers will carry an Android-based smartphone, which they are to use as their own for one month. After using the smartphone for two weeks, they will abstain from smoking for 48 hours. The phone will passively sense and record information from onboard sensors and send that information to a central server. When server based algorithms detect a pattern of signals likely associated with smoking behavior, the smoker will be queried regarding their current state (smoking?, not smoking but likely to in the next 10 minutes?, etc.). Likewise, when smokers are about to smoke but were not queried, they can indicate they are about to smoke. This information will be used to update algorithms using machine learning techniques. As such, in this study investigators will gain knowledge that will increase understanding of antecedents of smoking behavior and improve the accuracy with which smoking risk can be detected.

ELIGIBILITY:
Inclusion Criteria:

* generally healthy
* between the ages of 18 and 65
* smoking of at least 10 cig/day of a brand delivering ≥ 0.5 mg nicotine (FTC method) for > 1 year AND an afternoon expired CO concentration >5 ppm (to confirm inhalation) or morning urinary cotinine > 100 ng/mL
* willingness to carry and use a study smartphone as their own for one month

Exclusion Criteria:

* inability to attend all required sessions
* use of smokeless tobacco products
* current use of nicotine replacement therapy or other smoking cessation treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change in smoking behaviors as measured by an algorithm of social variables | up to 4 weeks
  phone calls (time, duration, coded identity of contact, including smoking status); SMS texting (time sent, coded identity of contact)

SECONDARY OUTCOMES:
Change in smoking behaviors as measured by an algorithm of motion variables | up to 4 weeks
  acceleration; direction and magnitude of gravity; device orientation
Change in smoking behaviors as measured by an algorithm of environmental variables | up to 4 weeks
  light; proximity; magnetic field; pressure; temperature
Change in smoking behaviors as measured by an algorithm of device interaction variables | up to 4 weeks
  running applications; applications installed; screen status
Change in smoking behaviors as measured by an algorithm of positioning variables | up to 4 weeks
  location; Bluetooth devices within range; available WiFi access points; ID for the current cell tower the device is connected to

CONTACTS AND LOCATIONS:
Overall Officials: Joseph McClernon, Ph.D, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States